CLINICAL TRIAL: NCT01301573
Title: Long Term Follow-Up Study for rAAV-GAD Treated Subjects
Status: Terminated | Type: Observational
Why Stopped: Due to financial reasons
Sponsor: Neurologix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GAD-LTFU
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- rAAV-GAD Treated Subjects: rAAV-GAD treated subjects who are being observed for long-term effects of the gene therapy product which they received from participating in a previous clinical study.
  Interventions: Biological: rAAV-GAD

INTERVENTIONS:
Biological: rAAV-GAD

SUMMARY:
The purpose of this observational study is the long term follow-up of Parkinson's patients who participated in a clinical trial in which they received AAV-GAD gene transfer into the subthalamic nucleus (STN) region of the brain. Patients will be followed once a year for up to five (5) years. The study will monitor and evaluate the long term effects of AAV-GAD and provide long term safety information.

ELIGIBILITY:
Inclusion Criteria:

* Participated in a clinical trial where they received AAV-GAD
* Able to give informed consent to participate in the study

Exclusion Criteria:

* Received Deep Brain Stimulation after receiving AAV-GAD
* Received any experimental device in the brain after receiving AAV-GAD
* Had any type of brain surgery after receiving AAV-GAD
* Received any experimental therapy (drug or biologic) for Parkinson's disease or any other indication after receiving AAV-GAD

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease patients who participated in a clinical trial in which they received AAV-GAD gene transfer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-01

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health Systems, Southfield, Michigan
  - Wake Forest University Health Science Center, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio